CLINICAL TRIAL: NCT01801774
Title: Quantitative Comparison of the Efficacy of Subtenon 20-mg Triamcinolone Injection With 0.1% Dexamethasone Eye Drop in Controlling Intraocular Inflammation After Phacoemulsification
Brief Title: Efficacy Comparison Study of Steroids to Control Post-operative Inflammation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Si234/2012
Record Dates: First submitted 2013-02-26; First posted 2013-03-01 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Inflammation; Intraocular Pressure
Keywords: post-operative inflammation; steroid; intraocular pressure
MeSH Terms: conditions — Inflammation | interventions — Triamcinolone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexamethasone (Placebo Comparator): Dexamethasone 0.1%/Tobramycin 0.3% eye drop 4 times per day for 28 days
  Interventions: Drug: Placebo
- Triamcinolone (Active Comparator): Subtenon 20-mg Triamcinolone injection
  Interventions: Drug: Subtenon 20-mg triamcinolone injection

INTERVENTIONS:
Drug: Subtenon 20-mg triamcinolone injection — Treatment arm will receive single subtenon 20-mg triamcinolone with gentamicin injection after uneventful phacoemulsification. 0.3% Tobramycin eye drop will be given to treatment arm for 28 days to blind the patient.
  Other Names: Triamcinolone
  Arms: Triamcinolone
Drug: Placebo
  Arms: Dexamethasone

SUMMARY:
Phacoemulsification is a quick method with less complication for cataract surgery. Due to the use of ultrasonic energy, it produced more post-operative inflammation than other methods. Many routes of steroid had been used to control post-operative inflammation. The investigators here compare the efficacy of single depot steroid subtenon injection (20-mg triamcinolone) with four-time-a-day steroid eye drop (0.1% dexamethasone) in controlling inflammation after uneventful phacoemulsification.

DETAILED DESCRIPTION:
Cataract is one of the most common causes of blindness in the world. Surgical removal of lens is the only treatment for cataract, which now shifts from extracapsular cataract extraction to phacoemulsification. Although phacoemulsification provides faster operating time and gives better optical result and rapid recovery to the patient, it causes more inflammation post-operatively compare with extracapsular cataract extraction. Corticosteroids eye drops are mainly use to control intraocular inflammation after the surgery.

Other routes of corticosteroids have been introduced to increase the intraocular level and to increase the patient's compliance. Subtenon triamcinolone injection is easy and safe. Antiinflammatory effect of single subtenon triamcinolone injection lasts about 4-6 weeks. This method has been used in combination with corticosteroid eye drop to control the inflammation after cataract surgery in uveitic patients. It shows potency in controlling of intraocular inflammation with lower rate of increasing the intraocular pressure. The investigators here quantitatively compare the efficacy of subtenon 20-mg triamcinolone injection with 0.1% dexamethasone eye drop in controlling intraocular inflammation after uneventful phacoemulsification.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18 years old
* Uncomplicated cataract patient scheduled for phacoemulsification and posterior chamber intraocular lens implantation
* No History of prior intraocular procedures or any eye diseases such as uveitis, glaucoma, diabetic retinopathy
* No History of systemic autoimmune diseases
* No History of allergy to corticosteroids or to any component of the study medications
* No History of using corticosteroids, non-steroidal anti-inflammatory drugs (NSAIDs), or immunomodulating agents within 3 months prior to surgery

Exclusion Criteria:

* Complications occurred during cataract surgery such as ruptured posterior capsule, vitreous loss, or dropped nucleus
* Pregnant and lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2012-05; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Anterior chamber reaction | postoperative day 28
  proportion of anterior chamber reaction grade 0 measured by anterior chamber inflammation score at postoperative day 28+/-5

SECONDARY OUTCOMES:
rate of increased intraocular pressure over 21 mmHg | preoperative, postoperative day 1,7,14,28,90
  rate of increased intraocular pressure over 21 mmHg by Goldman applanation tonometer
Changes of anterior chamber reaction over time | preoperative, postoperative day1, 7, 14, 28, 90
  repeated measure in changes of anterior chamber reaction over time from preoperative state to postoperative day 90

CONTACTS AND LOCATIONS:
Overall Officials: Pitipol Choopong, MD, Principal Investigator — Mahidol University
Locations (1):
- Siriraj Hospital, Bangkok Noi, Bangkok, Thailand